CLINICAL TRIAL: NCT01352273
Title: A Phase Ib Open-label Dose Escalation Study of MEK162 and RAF265 in Adult Patients With Advanced Solid Tumors Harboring RAS or BRAFV600E Mutations
Brief Title: MEK162 and RAF265 in Adult Patients With Advanced Solid Tumors Harboring RAS or BRAFV600E Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2102; 2010-023812-14 (EudraCT Number)
Record Dates: First submitted 2011-05-02; First posted 2011-05-11 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors
Keywords: advanced Solid tumors; harboring RAS; harboring BRAFV600E
MeSH Terms: interventions — binimetinib; RAF265

ARMS (1):
- MEK162 + RAF265 (Experimental)
  Interventions: Drug: MEK162 + RAF265

INTERVENTIONS:
Drug: MEK162 + RAF265

SUMMARY:
This is a multi- center, open-label, dose finding, Phase Ib study to be conducted in two stages: a dose escalation part to determine the maximum tolerated dose (MTD) safety and tolerability of concurrent administration of MEK162 and RAF265, followed by an expansion part to further assess the safety and preliminary anti-tumor efficacy of this oral combination within two separate patient populations: i) patients with advanced solid tumors harboring BRAFV600E mutations or ii) patients with advanced solid tumors harboring RAS mutations.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically or cytologically confirmed and non-resectable advanced solid tumors for which no further effective standard therapy exists.

* The patients' tumors must contain documented activating somatic BRAFV600E* , NRAS or KRAS mutations (except for pancreatic cancer)
* All patients enrolled MUST provide fresh or archival tumor samples at baseline to enable central confirmation of BRAF or KRAS/NRAS mutations
* Measurable, or non-measurable but evaluable disease as determined by RECIST
* Adequate bone marrow function
* Adequate hepatic and renal function
* Adequate cardiovascular function
* Negative serum β HCG test (female patients of childbearing potential only) within 72 hrs prior to first dose

Exclusion Criteria:

* Patients with a history of primary central nervous system tumors or brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases
* Current evidence of retinal disease; or ophthalmopathy as assessed by ophthalmologic examination at baseline that would be considered a risk factor for CSR/RVO (e.g., optic disc cupping, visual field defects, IOP > 21 mm Hg)
* Impaired cardio-/vascular function or clinically significant cardiovascular diseases, including any of the following:

  * History/evidence of acute coronary syndromes (including MI, unstable angina, CABG, coronary angioplasty, or stenting) ≤ 6 months prior to starting study drugs
  * Thromboembolic event (DVT, CVA, PE) ≤ 6 months prior to starting study
  * Symptomatic CHF, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality
  * Uncontrolled arterial hypertension, defined as BP > 140/100 mmHg (average of 3 consecutive readings)
* History of melena, hematemesis or hemoptysis within the last 3 months
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | during the first 28 days of treatment with RAF265 and MEK162

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events | 18 months
assess preliminary anti-tumor activity of the combination | every 8 weeks of treatment
  CT scan will be performed
Tumor skin and blood samples will be collected before and during treatment with RAF265 and MEK162 to assess the combination's effects on the RAF/MEK/MAPK pathway with the clinical outcomes | 18 months
Time versus plasma concentration profiles of RAF265 and MEK162 | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (3):
  - H. Lee Moffitt Cancer Center & Research Institute Moffitt 4, Tampa, Florida
  - Oregon Health & Science University OHSU 3, Portland, Oregon
  - University of Utah / Huntsman Cancer Institute Huntman 2, Salt Lake City, Utah
- Canada (2):
  - Pfizer Investigative Site, Edmonton, Alberta
  - Pfizer Investigative Site, Montreal, Quebec
- Pfizer Investigative Site, Oslo, Norway
- Pfizer Investigative Site, Madrid, Spain
- Pfizer Investigative Site, Zurich, Switzerland